CLINICAL TRIAL: NCT00863928
Title: Effects of Perioperative Belladonna and Opium Suppositories on Postoperative Pain and Morphine Consumption on Patients After Robotic Assisted Laparoscopic Radical Prostatectomy
Brief Title: Effects of Perioperative B&O Suppositories on Post-op Pain and Morphine Use After Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Principal Investigator, John Corman, MD, Principal Investigator, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB08100; IRB08100 (Other: Benaroya Research Institute)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Opium; Suppositories

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): No suppository given
- B & O suppository (Experimental): B & O suppository, belladonna 16.2 mg and opium 60 mg suppository (Paddock Laboratories, Minneapolis, MN)
  Interventions: Drug: belladonna 16.2 mg and opium 60 mg suppository

INTERVENTIONS:
Drug: belladonna 16.2 mg and opium 60 mg suppository — belladonna 16.2 mg and opium 60 mg suppository
  Other Names: B & O Suppository
  Arms: B & O suppository

SUMMARY:
This study is evaluating the effect of a Belladonna and Opium suppository administered intraoperatively on post operative pain after laparoscopic radical prostatectomy for prostate cancer. This is a blinded randomized study. 50% of patients will receive the suppository, 50% of patients will not. Neither you or your surgeon will know which group you are in.

DETAILED DESCRIPTION:
All patients undergoing LRP at Virginia Mason Medical Center between November 1, 2008 and July 30, 2009 were offered the opportunity to participate in a randomized double blind clinical trial. Operating surgeons were blinded to suppository placement which was administered after induction of anesthesia. All patients underwent a standardized anesthesia regimen. Post-operative pain was assessed by a visual analog scale (VAS) and post-operative narcotic use was calculated in intravenous morphine equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic radical prostatectomy at Virginia Mason, who do not have chronic pain or allergies to opioid analgesics are eligible for this study.

Exclusion Criteria:

* Women are excluded due to the absence of a prostate.
* Children are excluded due to the absence of prostate cancer in this group.
* Patients meeting any of the following will not be eligible for the study:

  * Patients at risk for complications from anticholinergic agents including those with a history of glaucoma, bronchial asthma, convulsive disorder, or high risk for delirium
  * History of previous allergies or adverse reactions to belladonna and opium and/or opioid analgesics
  * History of chronic pain or chronic use of opioid and nonopioid analgesics
  * History of alcohol or opioid dependency/abuse within last three months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Corman, MD, Principal Investigator — Benaroya Research Institute
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 1, 2008 through July 30, 2009. Subjects recruited at medical center
Groups:
- Control: no intervention
- B & O Suppository: belladonna 16.2 mg and opium 60 mg suppository
Period: Overall Study
Arm/Group | Control | B & O Suppository
Started | 94 | 41
Completed | 58 | 41
Not Completed | 36 | 0
Not completed — Protocol Violation | 26 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — surgery cancellation | 4 | 0
Not completed — medication allergy | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | B & O Suppository | Total
Number analyzed (Participants) | 94 | 41 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 20 | 68
  >=65 years | 46 | 21 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (6.86) | 62.7 (7) | 61.7 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 94 | 41 | 135
Region of Enrollment [Number; unit: participants]
  United States | 94 | 41 | 135

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment by Visual Analog Scale at Rest
Description: The Pain Assessment by Visual Analog Scale (VAS) consists of 100 millimeter (mm) horizontal line with two endpoints 1-100, labeled "no pain" and "worst possible pain. "No pain" is the minimum value and "worst possible pain" is the maximum value.
  Minimum value or "No Pain" is considered a better outcome.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Control | B & O Suppository
Number analyzed (Participants) | 94 | 41
millimeters | 19.08 (18) | 13.84 (9)

ADVERSE EVENTS:
Time Frame: 24 hours post-operatively
Description: Sedation, nausea, and pruritis will be assessed by nursing every 1 hour x 4 hours, then every 2 hours by 4, then every 4 hours up to 24 hours post-op
Arm/Group | Control | B & O Suppository
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/41
Other Adverse Events (participants affected / at risk) | 0/58 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes